CLINICAL TRIAL: NCT05821465
Title: Ambulatory Leadless Electrocardiogram Recorder Trial (ALERT Feasibility)
Brief Title: Ambulatory Leadless Electrocardiogram Recorder Trial Feasibility
Acronym: ALERT
Status: Completed | Type: Observational
Sponsor: HelpWear Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: V2.0
Record Dates: First submitted 2023-03-24; First posted 2023-04-20 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2023-04

CONDITIONS: Arrhythmias, Cardiac; Palpitation; Syncope; Light Headedness
MeSH Terms: conditions — Arrhythmias, Cardiac; Syncope; Dizziness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HeartWatch vs. Event Recorder: All patient-tagged (symptomatic) events recorded by the HeartWatch, and reference devices (Event Recorder) and all non-normal clinically significant rhythm auto-triggered and recorded events will be adjudicated and classified using literature-based definitions.
  Interventions: Device: HeartWatch
- HeartWatch vs. Holter: All patient-tagged (symptomatic) events recorded by the HeartWatch, and reference devices (Holter) and all non-normal clinically significant rhythm auto-triggered and recorded events will be adjudicated and classified using literature-based definitions.
  Interventions: Device: HeartWatch

INTERVENTIONS:
Device: HeartWatch — The HeartWatch monitoring device will be worn on the upper left arm for the same duration or up to 48 hours that the standard event recorder or holter monitor is worn. The subject will be provided with a HelpWear smartphone that is paired to the monitor and only used by the participant to tag any events that they may have during the Heartwatch monitoring session.

SUMMARY:
The goal of this study is to compare the heart signals that are received by a new heart monitoring device called the HeartWatch to heart signals that are recorded by existing monitors used in cardiology clinics today. The main question[s] it aims to answer are:

1. Does the HeartWatch recording allow characterization of tagged and abnormal arrhythmia events that are equivalent to the existing Event Recorder and Holter devices?
2. Does the HeartWatch recording allow for detection of QRS complexes that are equivalent to the predicate Holter lead I reference signal? Participants who have been recommended to receive a heart monitor for heart rhythm assessment will asked to wear the HeartWatch armband monitor at the same time as the standard heart monitor. They will be asked to flag symptoms (if they occur) on either the HeartWatch or on the Helpwear Smartphone. When their monitoring session for the standard heart monitor is complete, then the monitoring session for the HeartWatch armband is also complete.

DETAILED DESCRIPTION:
Two general types of consumer products are used to monitor patients with or at risk of heart rhythm disorders. Most estimate heart rhythm using blood flow (photoplethysmography) alone or in combination with activity sensors (accelerometer). These methods are not reliable in detecting heart rhythm abnormalities. Other methods record an ECG when the patient has symptoms. These devices are useful, but require the wearer to recognize their symptoms, attach the device and rest quietly to obtain an ECG recording of reasonable quality. The user then needs to send that information to a healthcare provider to verify. Hence, these consumer-based technologies are far from ideal. However, the diagnostic accuracy of single-lead ECG via wearable medical devices is excellent and, likely superior to a family physician's interpretation of a 12-lead ECG.3 High-quality ECG data from wearable devices that can unequivocally document AF can expedite its detection, allowing prompt diagnosis and appropriate prescription of antithrombotic and other therapies.

The HeartWatch arm band is designed to provide non-invasive, continuous single lead ECG data, irrespective of activity, the environment, and other factors. It continuously records ECG data for subsequent, offline analysis. The HeartWatch allows the user to note (flag) any symptoms they experience (e.g., palpitations, light-headedness, fainting, etc…) to allow for symptom-rhythm correlation and subsequent review by a physician. The HeartWatch displays all the elements of an ECG signal (i.e., PQRST) to facilitate diagnoses by physicians and is comparable to lead I of a traditional ECG system.

The HeartWatch is indicated for the extended diagnostic evaluation of patients with symptomatic and transient symptoms such as light-headedness, syncope and palpitations, as well as patients at risk for arrhythmias, but without significant symptoms.

The primary purpose of the study is to compare the interpretability of all tagged and all non-normal clinically significant arrhythmia events and the detection of QRS complexes by the HeartWatch, an upper armbased, ambulatory, single lead ECG collection tool, vs. conventional Event Recorder or Holter monitor reference device.

ELIGIBILITY:
Inclusion Criteria:

* At least 22 years of age at time of consent
* Clinically indicated for an Event Recorder or Holter
* Able to follow the protocol
* Provision of written-informed consent
* No functional implantable pacemaker or defibrillator
* Left bicep circumference > 22 cm and < 45 cm

Exclusion Criteria:

* Known allergy to any component of the Event Recorder
* Known allergy to any component of the Holter monitor
* Known allergy to any component of the HeartWatch
* Dextrocardia
* Implanted functional Pacemaker of Defibrillator
* Left bicep circumference < 22 cm
* Left bicep circumference > 45 cm

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients referred for extended ambulatory ECG monitoring will be approached for participation. A total of 150 subjects will be enrolled into the two parallel studies, 50 subjects in the HeartWatch vs Event recorder and 100 subjects in HeartWatch vs Holter monitor.
Sampling Method: Non-Probability Sample
Enrollment: 144 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-07-18 (Actual); Study Completion 2024-07-18 (Actual)

PRIMARY OUTCOMES:
HeartWatch arrhythmia event characterization accuracy | Events will be assessed for the duration of time each participants wears the HeartWatch and holter/event recorder, up to 48 hours.
  An arrhythmia diagnosis will be applied to all patient-tagged (symptomatic) events (HeartWatch, Event Recorder, and Holter) and all abnormal significant rhythm auto-triggered events (HeartWatch and Event Recorder) and recorded events (HeartWatch and Holter). For the HeartWatch to be considered comparable to the Holter and Event Recorder, the accuracy of the HeartWatch to categorize the correct arrhythmia must be > 85% of the combined Holter and Event Recorder data.
HeartWatch recording accuracy of QRS complexes | QRS complexes will be assessed for the duration of time each participants wears the HeartWatch and the holter monitor up to 48 hours.
  To be considered comparable to the Holter, the HeartWatch must detect > 90% of the QRS complexes recorded on the Holter lead I reference ECG signal

SECONDARY OUTCOMES:
Does the HeartWatch differ from the Event Recorder and Holter monitor in terms of adverse events? | Events will be assessed up to 48 hours of the patient wearing the HeartWatch.
  The incidence of adverse events will be collected and compared between the HeartWatch vs the standard heart monitors
Evaluate if the HeartWatch will be similarly preferred to the Event Recorder and Holter monitor. | Up to 48 hours
  Subjects will complete a questionnaire that will allow them to indicate their user preference on reture of the device.
The 10-minute averaged and paired PR/QRS intervals from the HeartWatch will be within 20 msec of the 10-minute averaged PR/QRS intervals from lead I of the Holter for at the same time points | Up to 48 hours.
  The 10-minute averaged PR, QRS, and QT intervals from the HeartWatch and Holter lead I will be analyzed using software created by HelpWear
the 10-minute averaged and paired QT intervals from the HeartWatch will be within 40 msec of the 10-minute averaged QT intervals from lead I of the Holter. | Up to 48 hours.
  The 10-minute averaged PR, QRS, and QT intervals from the HeartWatch and Holter lead I will be analyzed using software created by HelpWear

CONTACTS AND LOCATIONS:
Overall Officials: Derek Exner, MD, Study Director — HelpWear Inc.
Locations (1):
- Foothills Medical Centre, Calgary, Alberta, Canada